CLINICAL TRIAL: NCT06180798
Title: Cold Snare Endoscopic Mucosal Resection (C-EMR) Versus Hot Snare Endoscopic Mucosal Resection (H-EMR) for Large Colorectal Polyps (10-20 mm) - A Randomised Control Trail.
Brief Title: Cold Snare Endoscopic Mucosal Resection (C-EMR) Versus Hot Snare Endoscopic Mucosal Resection (H-EMR) for Large Colorectal Polyps (10-20 mm)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C-EMR VS H-EMR
Record Dates: First submitted 2023-10-21; First posted 2023-12-26 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Polyps of Colon; Polyps; Polyp Intestine
MeSH Terms: conditions — Colonic Polyps; Polyps; Intestinal Polyps

STUDY DESIGN:
Intervention Model Description: This is a single center randomized controlled study with two parallel groups with a 1:1 allocation ratio.
Who Masked: Participant
Masking Description: The patients will be randomised to C-EMR and H-EMR by a computer generated sequence provided in turn by the research assistant. The patient, pathologist and statistician will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cold snare endoscopic mucosal resection (C-EMR) (Active Comparator): All procedures will be performed by experienced endoscopists (>3 years of experience/>1000 polypectomies) with the patient in the left lateral position under propofol sedation.submucosal injection of saline mixed with methylene blue will be used (no epinephrine) followed by resection using snare without using electrocautery in C-EMR group.The polyp size will be assessed by boston biopsy forceps (open jaws -7mm) or boston jumbo biopsy forceps (open jaws 10mm) or submucosal injection needle (Olympus (4mm)). A standard snare will be used.After polypectomy, the area is inspected for residual polyp using NBI and if present, will be resected using biopsy forceps.
  Interventions: Procedure: cold snare endoscopic mucosal resection (C-EMR)
- Hot snare endoscopic mucosal resection (H-EMR) (Sham Comparator): All procedures will be performed by experienced endoscopists (>3 years of experience/>1000 polypectomies) with the patient in the left lateral position under propofol sedation.Using ERBE electrosurgical unit - EndoCut Q mode (effect interval duration) and forced coagulation mode in H-EMR group.The polyp size will be assessed by boston biopsy forceps (open jaws -7mm) or boston jumbo biopsy forceps (open jaws 10mm) or submucosal injection needle (Olympus (4mm)). A standard snare will be used.After polypectomy, the area is inspected for residual polyp using NBI and if present, will be resected using biopsy forceps.
  Interventions: Procedure: Hot snare endoscopic mucosal resection (H-EMR)

INTERVENTIONS:
Procedure: cold snare endoscopic mucosal resection (C-EMR) — All procedures will be performed by experienced endoscopists (>3 years of experience/>1000 polypectomies) with the patient in the left lateral position under propofol sedation.
  The polyp size will be assessed by boston biopsy forceps (open jaws -7mm) or boston jumbo biopsy forceps (open jaws 10mm) or submucosal injection needle (Olympus (4mm)). A standard snare will be used .
  submucosal injection of saline mixed with methylene blue will be used (no epinephrine) followed by resection using snare without using electrocautery in C-EMR group.After polypectomy, the area is inspected for residual polyp using NBI and if present, will be resected using biopsy forceps.
  Bleeding will be assessed for 2 mins to decide upon requirement of immediate hemostatic methods in the form of clipping or electrocoagulation.
  Arms: cold snare endoscopic mucosal resection (C-EMR)
Procedure: Hot snare endoscopic mucosal resection (H-EMR) — All procedures will be performed by experienced endoscopists (>3 years of experience/>1000 polypectomies) with the patient in the left lateral position under propofol sedation.
  The polyp size will be assessed by boston biopsy forceps (open jaws -7mm) or boston jumbo biopsy forceps (open jaws 10mm) or submucosal injection needle (Olympus (4mm)). A standard snare will be used.submucosal injection of saline mixed with methylene blue will be used.Using ERBE electrosurgical unit - EndoCut Q mode (effect interval duration) and forced coagulation mode in H-EMR group.
  After polypectomy, the area is inspected for residual polyp using NBI and if present, will be resected using biopsy forceps.
  Arms: Hot snare endoscopic mucosal resection (H-EMR)

SUMMARY:
OBJECTIVES The aim of the study is to compare the efficacy of cold snare EMR versus hot snare EMR for non-pedunculated polyps 10-20mm in size with respect to complete resection rates and adverse events.

DESIGN : A Randomised interventional study. Sample size: 330

DETAILED DESCRIPTION:
* This procedure will be performed by Endoscopists having above 3 years of experience you will be in the left lateral position under propofol sedation.
* In Both groups (a mixture of saline and blue dye will be injected beneath the surface layer,and then a snare(is a ring shaped device used to cut polyp after surrounding it- like a rubber band ) will be used to remove tissue without using heat in Cold Endoscopic mucosal resection group and using electrosurgical unit (to control bleeding and to rapidly dissect soft tissue in surgery) by EndoCut Q mode (ensures safe and effective removal of large lesions in particular large polyps) in Hot Endoscopic mucosal resection group.
* After polypectomy (the surgical removal of a polyp) the area is inspected for residual polyp (presence of any type of tissue) using NBI (Narrow band imaging) and if present, will be CUT OFF.

  * A Standard snare ( snare is a ring shaped device used to cut polyp after surrounding it- like a rubber band) is used to cut the polyps

ELIGIBILITY:
Inclusion Criteria:

* Adult above 18 years
* polyp size greater than 5-10mm.

Exclusion Criteria:

* Inflammatory bowel disease
* Familial Polyposis Syndromes
* Patient who is unable to understand study protocol or not consenting
* Severe coagulopathy (INR Greater than 1.5 platelets)
* Receiving antiplatelets withing 5 days of procedure
* If antiplatelets stopped for 5 days-they were restarted on next day after procedure.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Assess the complete resection rate | 1 YEAR
  Primary outcome will be tested with chi-square test or Fisher's exact test. The level of significance has been set at 5%. To quantify the magnitude of the difference the relative risk and odds ratio will be calculated with 95% confidence interval.

SECONDARY OUTCOMES:
Secondary outcomes include procedure time, cost and adverse events. | 1 YEAR
  Univariate and multivariate analysis will be done to determine which are the factors associated with clinical success and clinical recurrence. Kaplan-Meier survival analysis will be done for appearance clinical recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Krithi Krishna Koduri, MD, Principal Investigator — Asian Institute of Gastroenterology
Locations (1):
- Krithi Krishna Koduri, Hyderabad, Telanagana, India

IPD SHARING:
Plan to Share IPD: No